CLINICAL TRIAL: NCT00895440
Title: Neuropad Test for Detection of Sudomotor Dysfunction in Patients With Painful and Painless Diabetic Neuropathy and Charcot Neuroarthropathy
Brief Title: Role of Indicator Test (Neuropad) in Detecting Diabetic Neuropathy
Status: Completed | Type: Observational
Sponsor: Tameside Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Edward Jude, Consultant Physician, Tameside Hospital NHS Foundation Trust
Other Study IDs: Neuropad01
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetes; Diabetic neuropathy; neuropad; Painless peripheral diabetic neuropathy; Painful peripheral diabetic neuropathy; Autonomic peripheral neuropathy; Charcot neuroarthropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Diabetic patients without neuropathy
- 2: Diabetic patients with painless neuropathy
- 3: Diabetic patients with painful neuropathy
- 4: Diabetic patients with Charcot neuroarthropathy
- 5: Control non-diabetic subjects

SUMMARY:
Diabetes mellitus can result in damage to the nerves supplying the feet. Various tests can be used to assess nerve damage but no tests so far have been used to assess loss of sweating which can lead to dry skin, fissuring and ulceration. The indicator test (Neuropad) is a plaster which is applied to the sole of the feet just below the 1st and 2nd toes of both feet. If the color of the plaster changes to pink it indicates that there is no nerve damage to the nerves. However if the plaster retains the blue color or the color only partially changes to pink after 600 seconds then this is a positive test and the patient has nerve damage.

DETAILED DESCRIPTION:
With increasing nervous dysfunction, the function of the sweat glands in the feet also diminishes and can cease completely. As a result the skin becomes brittle and dry, making it more susceptible to fissuring and breakdown leading to foot ulceration. This is where the diagnosis using the Neuropad plaster might be useful. The Neuropad measures sweat production and have been proposed as a new test of neuropathy (8,9). The Neuropad examines the function of the sweat glands by means of a colour indicator. The indicator test enables the diagnosis of neuropathy in a substantial proportion of patients with normal clinical examination (10).

This colour indicator, a cobalt-II-salt, is applied in the form of a plaster to the area of skin on the patient's foot to be examined. In healthy subjects, the moisture (sweat) on the foot changes the colour of the Neuropad plaster from blue to pink normally within minutes. However, if the colour does not change completely or very slowly, this indicates initial nerve damage. This test is, as yet, the only one that examines changes in moistness of the foot. The speed and scale of the colour change of the Neuropad plaster can then be assessed as indicators of sudomotor function and thus as indicators of diabetic neuropathy as well. Although the test has been done in patients with diabetic neuropathy it has not been used as a discriminator in painless and painful neuropathy, or in patients with Charcot neuroarthropathy.

In this study we aim to assess the presence of sudomotor dysfunction in patients with painful and painless neuropathy and patients with Charcot foot.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or type 2 diabetes
2. Age 18-70 years
3. Presence of painless neuropathy
4. Presence of painful neuropathy
5. Presence of Charcot foot

Exclusion Criteria:

1. Patients with allergy to any metal
2. Peripheral vascular disease (defined as the absence of two or more foot pulses and an ankle brachial index of < 0.8)
3. Renal failure (serum creatinine > 130 micromol/l)
4. Foot ulceration or cellulitis or osteomyelitis
5. Patients taking drugs that affect sweating (corticosteroids, antihistamines, psychoactive drugs)
6. Chronic alcohol abuse
7. B12 deficiency (presence of anaemia, raised mean corpuscular volume, past history of abnormal B12 levels, treatment with B12)
8. Patients with any skin conditions affecting their feet(neurodermatitis, psoriasis, scleroderma, Raynaud syndrome, hyperhydrosis, acrocyanosis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 and type 2 diabetic patients with and without peripheral neuropathy (painless and painful) and Charcot neuroarthropathy; and non-diabetic subjects
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Identify patients with peripheral neuropathy with the Neuropad indicator test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jude, MD, MRCP, Principal Investigator — Tameside General Hospital
Locations (1):
- Tameside General Hospital, Ashton-under-Lyne, Lancashire, United Kingdom

REFERENCES:
- [Result] Papanas N, Papatheodorou K, Papazoglou D, Monastiriotis C, Christakidis D, Maltezos E. A comparison of the new indicator test for sudomotor function (Neuropad) with the vibration perception threshold and the clinical examination in the diagnosis of peripheral neuropathy in subjects with type 2 diabetes. Exp Clin Endocrinol Diabetes. 2008 Feb;116(2):135-8. doi: 10.1055/s-2007-984455. Epub 2007 Dec 20. PMID 18095233
- [Result] Papanas N, Papatheodorou K, Christakidis D, Papazoglou D, Giassakis G, Piperidou H, Monastiriotis C, Maltezos E. Evaluation of a new indicator test for sudomotor function (Neuropad) in the diagnosis of peripheral neuropathy in type 2 diabetic patients. Exp Clin Endocrinol Diabetes. 2005 Apr;113(4):195-8. doi: 10.1055/s-2005-837735. PMID 15891953